CLINICAL TRIAL: NCT00927199
Title: Efficacy of Consumption of High-oleic Canola and Flaxseed Oils in the Management of Hypercholesterolemia and Other Cardiovascular Risk Factors
Brief Title: Efficacy of High-oleic Canola and Flaxseed Oils for Hypercholesterolemia and Cardiovascular Disease Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canola Council of Canada (Other); Flax Canada 2015 Inc. (Industry); Agri-Food Research and Development Initiative (Unknown)
Responsible Party: Peter J.H. Jones, PhD; Principal Investigator, Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B2007:071
Record Dates: First submitted 2009-06-17; First posted 2009-06-24 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Disease
Keywords: High-Oleic Canola Oil; Flaxseed Oil; Monounsaturated Fatty Acids; Polyunsaturated Fatty Acids; Alpha Linolenic Acid; Cardiovascular; Hypercholesterolemia; Lipids; Inflammation; Metabolism
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-Oleic Canola Oil (Experimental)
  Interventions: Dietary Supplement: High-Oleic Canola Oil
- High-Oleic Canola/Flaxseed Oil Blend (Experimental)
  Interventions: Dietary Supplement: High-Oleic Canola/Flaxseed Oil Blend
- Western Diet (Active Comparator)
  Interventions: Dietary Supplement: Western Dietary Control

INTERVENTIONS:
Dietary Supplement: High-Oleic Canola Oil — Diets contained 35% energy as fat; of which 70% was provided by high-oleic canola oil (high in monounsaturated fat (oleic acid))
  Arms: High-Oleic Canola Oil
Dietary Supplement: High-Oleic Canola/Flaxseed Oil Blend — Diets contained 35% energy as fat; of which 70% was provided by a 1:1 blend of high-oleic canola oil and flaxseed oil (high in monounsaturated fat (oleic acid) and omega-3 polyunsaturated fat (alpha-linolenic acid))
  Arms: High-Oleic Canola/Flaxseed Oil Blend
Dietary Supplement: Western Dietary Control — Diets contained 35% energy as fat; of which 70% was provided by a blend of oils typical to the Western diet (high in saturated fat and omega-6 polyunsaturated fat (linoleic acid))
  Arms: Western Diet

SUMMARY:
The purpose of this study is to assess the efficacy of high-oleic canola oil and a high-oleic canola/flaxseed oil blend as compared to a typical Western diet on plasma lipids, fatty acid profiles, and risk factors associated with cardiovascular disease in hypercholesterolemic patients. Furthermore, the metabolism of dietary oleic acid and alpha-linolenic acid contained in high-oleic canola oil and flaxseed oil will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Fasting serum LDL-Cholesterol >3.0 mmol/L
* Body mass index (BMI) between 22-36 kg/m2

Exclusion Criteria:

* smoking
* use of lipid lowering therapy
* documented cardiovascular/atherosclerotic disease
* inflammatory disease
* diabetes
* uncontrolled hypertension
* kidney disease
* other systemic diseases
* cancer
* chronic alcohol consumption (> 2 servings/day)
* excessive exercise expenditure (> 4000 kcal/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Serum Lipids | Baseline (Day 1,2) and Endpoint (Day 28,29) of each experimental phase
Inflammatory Biomarkers: C-Reactive Protein, Interleukin-6, sE-Selectin, sVCAM-1, sICAM-1 | Study Baseline (Day 1,2) and Endpoint (Day 28,29) of each experimental phase
Intima-Medial Thickness by Carotid Ultrasound | Study Baseline (during Day 1-3) and Endpoint (during Day 24-26) of each experimental phase
Energy Expenditure by Indirect Calorimetry | Study Baseline (during Week 1) and Endpoint (during Week 4) of each experimental phase
Body Composition by Dual Emission X-Ray Absorptiometry (DEXA) | Baseline (Day1,2) and Endpoint (Day 28,29) of each experimental phase
Oxidation and Conversion of U-13C-Alpha Linolenic Acid | Day 27 (time 0-8 hrs), Day 28 (24 hrs), Day 29 (48 hrs) of each experimental phase
Plasma Fatty Acid Concentrations | Baseline (Day 1,2) and Endpoint (Day 28,29) of each experimental phase

SECONDARY OUTCOMES:
Arterial Stiffness Index by Pulse Wave Analysis | Baseline (Day 1,2) and Endpoint (Day 28,29) of each experimental phase

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba - Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Gillingham LG, Harris-Janz S, Jones PJ. Dietary monounsaturated fatty acids are protective against metabolic syndrome and cardiovascular disease risk factors. Lipids. 2011 Mar;46(3):209-28. doi: 10.1007/s11745-010-3524-y. Epub 2011 Feb 10. PMID 21308420
- [Result] Gillingham LG, Harding SV, Rideout TC, Yurkova N, Cunnane SC, Eck PK, Jones PJ. Dietary oils and FADS1-FADS2 genetic variants modulate [13C]alpha-linolenic acid metabolism and plasma fatty acid composition. Am J Clin Nutr. 2013 Jan;97(1):195-207. doi: 10.3945/ajcn.112.043117. Epub 2012 Dec 5. PMID 23221573
- [Result] Gillingham LG, Robinson KS, Jones PJ. Effect of high-oleic canola and flaxseed oils on energy expenditure and body composition in hypercholesterolemic subjects. Metabolism. 2012 Nov;61(11):1598-605. doi: 10.1016/j.metabol.2012.04.016. Epub 2012 Jun 12. PMID 22698766
- [Result] Gillingham LG, Gustafson JA, Han SY, Jassal DS, Jones PJ. High-oleic rapeseed (canola) and flaxseed oils modulate serum lipids and inflammatory biomarkers in hypercholesterolaemic subjects. Br J Nutr. 2011 Feb;105(3):417-27. doi: 10.1017/S0007114510003697. Epub 2010 Sep 29. PMID 20875216
- [Derived] Jones PJ, Lin L, Gillingham LG, Yang H, Omar JM. Modulation of plasma N-acylethanolamine levels and physiological parameters by dietary fatty acid composition in humans. J Lipid Res. 2014 Dec;55(12):2655-64. doi: 10.1194/jlr.P051235. Epub 2014 Sep 28. PMID 25262934